CLINICAL TRIAL: NCT01474746
Title: A Controlled Trial of Sertraline in Young Children With Fragile X Syndrome
Brief Title: Trial of Sertraline to Treat Children With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Randi J. Hagerman, MD (Other)
Responsible Party: Sponsor-Investigator, Randi J. Hagerman, MD, Principle Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 271070; R40MC22641 (Other Grant/Funding Number: Health Resources and Services Administration (HRSA))
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Pediatrics; sertraline; autism
MeSH Terms: conditions — Fragile X Syndrome; Autistic Disorder | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): This arm will undergo identical treatment and assessments as the experimental group, with the exception of the active agent, sertraline. This group will be placed on a placebo.
  Interventions: Drug: Placebo
- Active (Experimental): This arm will undergo identical treatment and assessments as the placebo group. This group will receive the active agent, sertraline.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Liquid sertraline (20 mg/mL) will be dosed in an age-dependent manner. Participants aged 2-3 years of age will be given 2.5 mg (0.125 mL) of liquid sertraline once per day for a period of six months. Participants aged 4 years to 5 years 8 months will be given 5 mg (0.25 mL) of liquid sertraline once per day for a period of six months.
  Other Names: Zoloft
  Arms: Active
Drug: Placebo — The placebo will be dosed in an age-dependent manner. Participants aged 2-3 years of age will be given 2.5 mg (0.125 mL) of liquid placebo once per day for a period of six months. Participants aged 4 years to 5 years 8 months will be given 5 mg (0.25 mL) of liquid placebo once per day for a period of six months.
  Arms: Placebo

SUMMARY:
This study is a control trial of sertraline (Zoloft) in fragile X syndrome children aged 2 years to 5 years 8 months old. The trial is six months long, and each participant will receive a series of tests at both the beginning and end of the study. The researchers hope to show improvements in language and a decrease in autistic symptoms.

DETAILED DESCRIPTION:
This is a single center study and the UC Davis MIND Institute for fragile X syndrome (FXS) patients aged between 2 years and 5 years, 8 months old funded by the Health Resources and Services Administration (HRSA). It is a double-blind control trial of sertraline (Zoloft), an anti-depressant typically used in the treatment of depression, obsessive-compulsive disorder, panic disorder, and other conditions. The researchers are investigating the use of this selective serotonin reuptake inhibitor (SSRI) in FXS because a retrospective study has shown significant improvements in language and decreases in autistic behavior. There is also emerging evidence regarding the stimulation of brain-derived neurotrophic factor (BDNF) and the stimulation of neurogenesis when an SSRI is given early on in the development of animal models of Down syndrome. The researchers hope to see improvements in language stimulation, social gaze and social reciprocity, spatial attention, and a decrease in autistic behaviors.

The aim of this study is to carry out a double-blind placebo controlled trial of sertraline in children with FXS who are between the ages of 2 years and 5 years, 8 months old. At baseline, the researchers will assess behavioral and cognitive development. These children will be treated for six months with either sertraline or placebo. At the end of the six months, the researchers assess the same behavioral and cognitive measures as at the beginning of the study. The researchers will also assess the side effects of the sertraline treatment throughout the study.

On March 14, 2017 two secondary outcomes for each of the primary outcomes were added for clarification of measurements at baseline visit and at six-month visit. In April 2017 additional updates were made to report primary and secondary outcome results. By June 2, 2017 all outstanding secondary outcome results had been added.

In July 2017, additional updates to the outcome measures and limitations sections were made to address PRS review comments. In the process of responding to these comments, a duplicate reported outcome measure was identified and deleted.

In August 2017, additional updates to the outcome measures were made to address PRS review comments issued in response to the July 2017 updates.

ELIGIBILITY:
Inclusion Criteria:

* Fragile X Syndrome

Exclusion Criteria:

* Current or past SSRI treatment
* Current or past MAOI (monoamine oxidase inhibitor ) treatment
* Serious co-morbid medical disorder affecting brain function and behavior (not including fragile X syndrome).
* Uncontrolled seizure disorder or epilepsy
* Bipolar disorder
* Latex allergies

Ages: 24 Months to 68 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Hagerman, MD, Principal Investigator — UC Davis MIND Institute; Kathleen Angkustsiri, MD, Principal Investigator — UC Davis MIND Institute
Locations (1):
- UC Davis M.I.N.D. Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Active
Started | 30 | 27
Completed | 27 | 25
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 27 | 57
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 27 | 21 | 48
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Mullen Scales of Early Learning - Expressive Language Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the baseline and 6-month follow-up raw scores from the expressive language scale. This scale's raw scores range from 0 to 50. The lower the score on this scale, the weaker the ability; the higher the score, the greater the ability. The MSEL was administered at the baseline visit and at the 6-month follow-up visit.
Time Frame: From baseline visit to six-month visit.
Population: Two subjects from the sertraline arm discontinued - 1 lost to follow up, 1 withdrew consent Three subjects from the placebo arm discontinued - 1 lost to follow up, 2 withdrew consent
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
units on a scale
  Baseline | 19.3 (9.68) | 21.3 (10.32)
  Follow-Up | 21.3 (9.59) | 25.04 (10.78)

2. Primary Outcome: Clinical Global Impression - Improvement
Description: The Clinical Global Impression - Improvement (CGI-I) is used to measure the overall behavioral change of an individual and their therapeutic response. The CGI-I is a 3-item observer-rated scale administered by the physician to the caregiver, who assesses improvement using a 7-point scale: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse. Therefore, the lower the score, the greater the behavioral improvement as rated by the caregiver. Shown here are the CGI-I mean scores from the 6-month follow-up visit.
Time Frame: 6-month follow-up visit score
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
units on a scale | 2.59 (0.84) | 2.28 (1.06)

3. Primary Outcome: Change in Mullen Scales of Early Learning - Expressive Language Standard T Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language and expressive language. Based on the raw score obtained by the participant in each scale the scoring software computes T scores, percentile ranks, and age equivalents for each scale separately. Shown here are the baseline and 6-month follow-up T scores from the expressive language scale. T scores have a range of 20 to 80, a mean of 50, and a standard deviation of 10. Any child scoring at or below 1.5 standard deviations below the average is considered presenting significant delays. The lower the T score, the worse the outcome. The MSEL was administered at the baseline visit and at the 6-month follow-up visit.
Time Frame: From baseline visit to six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
T scores
  Baseline | 23.3 (5.8) | 25.8 (11.78)
  6-Month Follow-Up | 22.6 (6.47) | 25.8 (10.87)

4. Secondary Outcome: Autism Diagnostic Observation Schedule
Description: The Autism Diagnostic Observation Schedule (ADOS-2) assesses and diagnoses autism spectrum disorder. This test was administered at baseline and at the six-month follow-up visit. The choice to administer Module 1 or Module 2 depends on the verbal ability of each subject: Module 1 is used for children who are 31 months and older and/or who do not consistently use phrase speech, and Module 2 is used for children of any age who use phrase speech but are not verbally fluent. The scoring algorithm gives an overall total, which ranges from 0 to 28. The higher the score, the higher the level of autism-related symptoms. The overall total ranges from 0 to 28. On Module 1, for children with few to no words, scores at 11 and above indicate autism spectrum; for children with some words, the cutoff is scores 8 and above. On Module 2, the cutoff for autism spectrum is 7 or above for kids under 5 years, and 8 or above for those 5 years and older.
Time Frame: At baseline visit
Population: The ADOS was not administered to all subjects at baseline due to the PI's decision to remove this assessment from the protocol partway through the study; due to staff oversight, however, this assessment remained listed among the measures in the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 24
units on a scale | 10.73 (6.23) | 11.00 (6.57)

5. Secondary Outcome: Visual Analog Scale
Description: The Visual Analog Scale will be used to measure the severity of three specific behavioral symptoms chosen by the caregiver(s). Parents mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. The parents choose two key behaviors that they want to target for this trial (e.g., aggression, hyperarousal, anxiety, hyperactivity) and the third target measurement is language/communication. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 6-month visit. The calculated distance in cm between the baseline and 6-month visit marks thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side, at baseline. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
centimeters | 2.95 (1.72) | 2.62 (1.74)

6. Secondary Outcome: Eye Tracking
Description: There are several eye tracking measures, each intended to measure different outcomes including social gaze, social reciprocity, and attention. All stimuli are presented on a Tobii T120 binocular eye tracker monitor. The system consists of a high-resolution camera embedded in a 17-inch TFT monitor. Stimuli consist of sixty colored photographs of adult human face (equal numbers of males and females, different races and ethnicities) from the NimStim Face Stimulus Set, each showing a calm, happy, or fearful expression, and sixty scrambled versions of the face images. Shown here are the averaged response times (in seconds) to the presented stimuli, at the baseline visit.
Time Frame: At baseline visit
Population: Data were collected and analyzed on those participants who were compliant with the eye tracking protocol: 13 in the placebo group, and 9 in the active group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Active
Number analyzed (Participants) | 13 | 9
seconds | 0.510136154 (0.056) | 0.451205556 (0.07)

7. Secondary Outcome: Preschool Language Scale-fifth Edition (PLS-5): AC+EC Total Raw Score
Description: The Preschool Language Scale-fifth edition (PLS-5) is designed to measure auditory comprehension (AC) and expressive communication (EC) for children birth to 7 years 11 months. The measure examines the child's attention, play, gestures, social communication, semantics, language structure, integrative language skills and emergent literacy skills. The PLS-5 has expanded coverage of early play behaviors, concepts, Theory of Mind, as well as emergent literacy skills. The PLS-5 yields norm-referenced scores including standard scores, percentile ranks and age equivalents for the AC and EC scales as well as for Total Language (TL). Raw score ranges are 0 to 65 in AC, 0 to 67 in EC, and therefore 0 to 132 in TL (calculated by summing AC+EC raw scores). The higher the scores, the greater the language ability. Shown here are the mean TL raw scores from the baseline visit.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
units on a scale | 53.90 (18.84) | 55.59 (21.13)

8. Secondary Outcome: Sensory Processing Measure - Preschool (SPM-P) Social Participation: Raw Score
Description: The Sensory Processing Measure - Preschool (SPM-P) is a questionnaire that was used to measure specific problems, including under- and over-responsiveness, sensory-seeking behavior, and perceptual problems in multiple environments (at home, at school, and in the community) for children aged 2 to 5 years old. The SPM-P provides norm-referenced standard scores for two higher level integrative functions (praxis and social participation) and five sensor sensory systems (visual, auditory, tactile, proprioceptive, and vestibular functioning). Reported here is the Social Participation subscale mean raw score, which ranges from 8 to 32. The lower the raw score, the more limited the child's level of social participation. The higher the score, the greater the child's level of social participation.
Time Frame: At baseline visit
Population: The SPM-P was removed from the protocol after the trial was initiated and was therefore not administered to 1 subject in the active treatment group at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 26
units on a scale | 20.6 (6.85) | 20.5 (5.49)

9. Secondary Outcome: Sensory Profile - Sensation Seeking Subscale Raw Score
Description: The Sensory Profile is designed to measure sensory-related difficulties. This measure will be administered to the primary caregiver of each subject to measure the caregiver's sensory ability and its impact on the subject. Of the four subscales scored in the Sensory Profile, the "Sensation Seeking" subscale mean raw scores for the placebo and treatment groups are reported here. This subscale has a raw scores range from 0 to 95, with scores 0-6 indicating that the child is sensation seeking much less than others, 7-19 less than others, 20-47 just like the majority of others, 48-60 more than others, and 61-95 much more than others.
Time Frame: At baseline visit
Population: The Sensory Profile was not administered to all subjects at baseline due to the PI's decision to remove this assessment from the protocol partway through the study; due to staff oversight, however, this assessment remained listed among the measures in the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 22 | 18
units on a scale | 47.86364 (7.97195) | 47.83333 (7.69454)

10. Secondary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) - Adaptive Behavior Composite Standard Score
Description: The Vineland-II measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Vineland-II is a survey that is administered to a parent or caregiver using a semi-structured interview format and is organized around four Behavior Domains: Communication, Daily Living Skills, Socialization, and Motor Skills. Each subtest is scored with a standard score X=100 ± 15 and summed to calculate the Adaptive Behavior Composite (ABC) using age-adjusted scoring tables. Reported here are the ABC mean standard scores for the placebo and treatment groups baseline. The ABC ranges from 20 to 160 and indicates low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Time Frame: At baseline visit
Population: This assessment was introduced to the protocol partway through the study, and therefore there were only 20 subjects (10 placebo and 10 active) who were administered the Vineland-II at both their baseline and follow-up visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 10 | 10
units on a scale | 73.3 (10.08905) | 66.5 (16.84076)

11. Secondary Outcome: Mullen Scales of Early Learning - Visual Reception Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean baseline raw scores from the Visual Reception scale. This scale's raw scores range from 0 to 50. The lower the score on this scale, the weaker the child's ability for visual reception; the higher the score, the greater the ability for visual reception.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
units on a scale | 28.9 (7.94) | 26.3 (9.50)

12. Secondary Outcome: Mullen Scales of Early Learning - Fine Motor Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean raw scores from the Fine Motor scale at the baseline visit. This scale's raw scores range from 0 to 49. The lower the score on this scale, the weaker the child's fine motor skills; the higher the score, the greater the child's fine motor skills.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
units on a scale | 24.8 (5.26) | 23.1 (7.13)

13. Secondary Outcome: The Autism Diagnostic Observation Schedule (ADOS-2)
Description: as for outcome 4
Time Frame: At six month visit
Population: The ADOS was not administered to all subjects at the six-month visit due to the PI's decision to remove this assessment from the protocol partway through the study; due to staff oversight, however, the ADOS remained listed in the protocol. Also, 2 sertraline and 3 placebo subjects discontinued and were thus administered no follow-up ADOS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 26 | 24
units on a scale | 11.00 (5.31) | 11.67 (6.59)

14. Secondary Outcome: The Visual Analog Scale
Description: The Visual Analog Scale will be used to measure the severity of three specific behavioral symptoms chosen by the caregiver(s). Parents mark on a visual line measuring 10 cm with "worst behavior" at 0 cm and "best behavior" at 10 cm. The parents choose two key behaviors that they want to target for this trial (e.g., aggression, hyperarousal, anxiety, hyperactivity) and the third target measurement is language/communication. For each behavior the caregiver is instructed to mark their impression of the behavior at baseline visit and again at the 6-month visit. The calculated distance in cm between the baseline and 6-month visit marks thereby demonstrates whether each behavior improved, worsened, or stayed the same during the study, and by how much. Shown here is the mean distance in cm from the "worst behavior" side, at the 6-month visit. The smaller the value, the worse the behavior. The range is minimum 0 cm to maximum 10 cm.
Time Frame: At six-month visit
Population: Two subjects from the sertraline arm discontinued - 1 lost to follow up, 1 withdrew consent. An additional subject from the sertraline arm was not administered this measure at the 6-month visit due to staff oversight.
  Three subjects from the placebo arm discontinued - 1 lost to follow up, 2 withdrew consent
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 24
units on a scale | 5.16 (2.03) | 5.58 (2.58)

15. Secondary Outcome: Eye Tracking
Description: There are several eye tracking measures, each intended to measure different outcomes including social gaze, social reciprocity, and attention. All stimuli are presented on a Tobii T120 binocular eye tracker monitor. The system consists of a high-resolution camera embedded in a 17-inch TFT monitor. Stimuli consist of sixty colored photographs of adult human face (equal numbers of males and females, different races and ethnicities) from the NimStim Face Stimulus Set, each showing a calm, happy, or fearful expression, and sixty scrambled versions of the face images. Shown here are the averaged response times (in seconds) to the presented stimuli, at the 6-month follow-up visit.
Time Frame: At six-month visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Active
Number analyzed (Participants) | 13 | 9
seconds | 0.505969231 (0.08) | 0.538312222 (0.095)

16. Secondary Outcome: Preschool Language Scale-fifth Edition (PLS-5): AC+EC Total Raw Score
Description: The Preschool Language Scale-fifth edition (PLS-5) is designed to measure auditory comprehension (AC) and expressive communication (EC) for children birth to 7 years 11 months. The measure examines the child's attention, play, gestures, social communication, semantics, language structure, integrative language skills and emergent literacy skills. The PLS-5 has expanded coverage of early play behaviors, concepts, Theory of Mind, as well as emergent literacy skills. The PLS-5 yields norm-referenced scores including standard scores, percentile ranks and age equivalents for the AC and EC scales as well as for Total Language (TL). Raw score ranges are 0 to 65 in AC, 0 to 67 in EC, and therefore 0 to 132 in TL (calculated by summing AC+EC raw scores). The higher the scores, the greater the language ability. Shown here are the mean TL raw scores from the 6-month follow-up visit.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
units on a scale | 59.89 (18.11) | 62.80 (21.70)

17. Secondary Outcome: Sensory Processing Measure-Preschool (SPM-P) Social Participation: Raw Score
Description: The Sensory Processing Measure - Preschool (SPM-P) is a questionnaire that was used to measure specific problems, including under- and over-responsiveness, sensory-seeking behavior, and perceptual problems in multiple environments (at home, at school, and in the community) for children aged 2 to 5 years old. The SPM-P provides norm-referenced standard scores for two higher level integrative functions (praxis and social participation) and five sensor sensory systems (visual, auditory, tactile, proprioceptive, and vestibular functioning). The SPM-P was administered to the caregiver at baseline and again at the 6-month follow-up visit. Reported here is the Social Participation subscale mean raw score from the 6-month visit, which ranges from 8 to 32. The lower the raw score, the more limited the child's level of social participation. The higher the score, the greater the child's level of social participation.
Time Frame: At six-month visit
Population: 2 subjects from the sertraline arm discontinued - 1 lost to follow up, 1 withdrew consent. 3 subjects from the placebo arm discontinued - 1 lost to follow up, 2 withdrew consent. The SPM-P was removed from the protocol after the trial was initiated and was therefore not administered to 4 placebo and 3 treatment recipients at the 6-month visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 23 | 22
units on a scale | 19.7 (6.41) | 18.0 (6.23)

18. Secondary Outcome: Sensory Profile - Sensation Seeking Subscale Raw Score
Description: as for outcome 9
Time Frame: At six-month visit
Population: The Sensory Profile assessment was not administered to any subjects at the follow-up visit due to revisions to the protocol.
Arm/Group | Placebo | Active
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) Adaptive Behavior Composite Standard Score
Description: The Vineland-II measures the personal and social skills of individuals from birth through adulthood. It was designed to assess handicapped and non-handicapped persons in their personal and social functioning and is appropriate for individuals of all ages. The Vineland-II is a survey that is administered to a parent or caregiver using a semi-structured interview format and is organized around four Behavior Domains: Communication, Daily Living Skills, Socialization, and Motor Skills. Each subtest is scored with a standard score X=100 ± 15 and summed to calculate the Adaptive Behavior Composite (ABC) using age-adjusted scoring tables. Reported here are the ABC mean standard scores for the placebo and treatment groups at the 6-month visit. The ABC ranges from 20 to 160 and indicates low (20-70), moderately low (70-85), adequate (85-115), moderately high (115-130), or high (130-160) overall adaptive functioning.
Time Frame: At six-month visit
Population: This assessment was only introduced to the protocol partway through the trial. As such, only 20 subjects (10 placebo, 10 active) were administered the Vineland-2 at both baseline and follow-up visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 10 | 10
units on a scale | 74.5 (7.50185) | 66.4 (17.68364)

20. Secondary Outcome: Mullen Scales of Early Learning - Visual Reception Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean raw scores from the Visual Reception scale at the 6-month follow-up visit. This scale's raw scores range from 0 to 50. The lower the score on this scale, the weaker the child's ability for visual reception; the higher the score, the greater the ability for visual reception.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
units on a scale | 30.9 (6.73) | 32.4 (10.46)

21. Secondary Outcome: Mullen Scales of Early Learning - Visual Reception Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean baseline age-equivalent scores from the Visual Reception scale. This scale's age-equivalent scores for each of the five scales are calculated from the raw scores for each scale, using the MSEL Age Equivalents table. Age-equivalent scores for each scale range from 0 to 70 months, with lower scores indicating that a child's visual reception is at a level typical of younger ages, and higher scores indicating that a child's visual reception is at a level typical of older ages.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
months | 28.2 (10.53) | 25.3 (11.59)

22. Secondary Outcome: Mullen Scales of Early Learning - Visual Reception Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean age-equivalent scores from the Visual Reception scale at the 6-month follow-up visit. This scale's age-equivalent scores for each of the five scales are calculated from the raw scores for each scale, using the MSEL Age Equivalents table. Age-equivalent scores for each scale range from 0 to 70 months, with lower scores indicating that a child's visual reception is at a level typical of younger ages, and higher scores indicating that a child's visual reception is at a level typical of older ages.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
months | 30.6 (9.60) | 33.7 (15.06)

23. Secondary Outcome: Mullen Scales of Early Learning - Fine Motor Raw Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean raw scores from the Fine Motor scale at the 6-month follow-up visit. This scale's raw scores range from 0 to 49. The lower the score on this scale, the weaker the child's fine motor skills; the higher the score, the greater the child's fine motor skills.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
units on a scale | 25.2 (4.96) | 27.3 (8.06)

24. Secondary Outcome: Mullen Scales of Early Learning - Fine Motor Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean baseline age-equivalent scores from the Fine Motor scale. This scale's age-equivalent scores for each of the five scales are calculated from the raw scores for each scale, using the MSEL Age Equivalents table. Age-equivalent scores for each scale range from 0 to 70 months, with lower scores indicating that a child's fine motor skills are at a level typical of younger ages, and higher scores indicating that a child's fine motor skills are at a level typical of older ages.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
months | 24.5 (6.97) | 22.7 (8.66)

25. Secondary Outcome: Mullen Scales of Early Learning - Fine Motor Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. Shown here are the mean age-equivalent scores from the Fine Motor scale at the 6-month follow-up visit. This scale's age-equivalent scores for each of the five scales are calculated from the raw scores for each scale, using the MSEL Age Equivalents table. Age-equivalent scores for each scale range from 0 to 70 months, with lower scores indicating that a child's fine motor skills are at a level typical of younger ages, and higher scores indicating that a child's fine motor skills are at a level typical of older ages.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
months | 25.0 (6.91) | 28.4 (10.91)

26. Secondary Outcome: Mullen Scales of Early Learning - Cognitive T Score Sum
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor (not administered because it was out of age range for most subjects), visual reception, fine motor, receptive language and expressive language. Based on the raw score obtained by the participant in each scale, the scoring software computes T scores for each scale separately. Each scale's T score has a range of 20 to 80, a mean of 50, and a standard deviation of 10, and the lower the T score, the lower the child's cognitive and developmental ability. Cognitive T score sum is the sum of the T scores for each scale administered; since 4 scales were administered, the sum's range is 80 to 320, with lower sums indicating lower overall ability. The MSEL was administered at the baseline visit and at the 6-month follow-up visit, and mean baseline cognitive T score sums for the placebo and treatment groups are shown here.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
T scores | 96.0 (21.97) | 99.7 (33.46)

27. Secondary Outcome: Mullen Scales of Early Learning - Cognitive T Score Sum
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor (not administered because it was out of age range for most subjects), visual reception, fine motor, receptive language and expressive language. Based on the raw score obtained by the participant in each scale, the scoring software computes T scores for each scale separately. Each scale's T score has a range of 20 to 80, a mean of 50, and a standard deviation of 10, and the lower the T score, the lower the child's cognitive and developmental ability. Cognitive T score sum is the sum of the T scores for each scale administered; since 4 scales were administered, the sum's range is 80 to 320, with lower sums indicating lower overall ability. The MSEL was administered at the baseline and 6-month follow-up visits, and mean cognitive T score sums from the 6-month follow-up visit for the placebo and treatment groups are shown here.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
T scores | 93.0 (20.33) | 105.4 (40.27)

28. Secondary Outcome: Mullen Scales of Early Learning - Summary Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language and expressive language. Based on the raw score obtained by the participant in each scale, the scoring software computes T scores, percentile ranks, and age equivalents for each scale separately, as well as a cognitive T score sum and summary age-equivalent score to characterize overall early developmental ability. Summary age-equivalent scores range from 0 to 70 months, with lower scores indicating that a child's ability is at a level typical of younger ages, and higher scores indicating that a child's ability is at a level typical of older ages. The MSEL was administered at the baseline visit and at the 6-month follow-up visit, and mean baseline summary age-equivalent scores for the placebo and treatment groups are shown here.
Time Frame: At baseline visit
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 30 | 27
months | 24.8 (9.33) | 26.8 (8.89)

29. Secondary Outcome: Mullen Scales of Early Learning - Summary Age-equivalent Score
Description: The Mullen Scales of Early Learning (MSEL) is a cognitive test to measure cognitive ability and language development. The test has five scales: gross motor, visual reception, fine motor, receptive language and expressive language. Based on the raw score obtained by the participant in each scale, the scoring software computes T scores, percentile ranks, and age equivalents for each scale separately, as well as a cognitive T score sum and summary age-equivalent score to characterize overall early developmental ability. Summary age-equivalent scores range from 0 to 70 months, with lower scores indicating that a child's ability is at a level typical of younger ages, and higher scores indicating that a child's ability is at a level typical of older ages. The MSEL was administered at the baseline visit and at the 6-month follow-up visit, and mean summary age-equivalent scores at the 6-month follow-up visit for the placebo and treatment groups are shown here.
Time Frame: At six-month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Placebo | Active
Number analyzed (Participants) | 27 | 25
months | 23.6 (10.76) | 30.1 (12.64)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected via non-systematic assessment (based on parent/caregiver reporting) throughout the 6-month period of each subject's participation in the study, as well as via systematic assessment (physical exams) at the baseline, 3-month, and 6-month timepoints.
Arm/Group | Placebo | Active
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 26/30 | 25/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | Active (N=27)
Tantrums (Psychiatric disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Self-injurious behavior (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Hand flapping (Psychiatric disorders) | 1 (1) | 0 (0)
Genital infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Decreased verbalization (General disorders) | 1 (1) | 0 (0)
Deciduous teeth eruption (General disorders) | 1 (1) | 0 (0)
Bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal Electroencephalogram (Investigations) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Falling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drooling (General disorders) | 1 (1) | 1 (1)
Dilated pupils (Eye disorders) | 1 (1) | 0 (0)
Biting clothing (General disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disturbance (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 1 (2)
Loss of appetite (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Sweating (Endocrine disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Bruxism (General disorders) | 0 (0) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 5 (8) | 3 (5)
Hyperactivity (Psychiatric disorders) | 4 (4) | 3 (4)
Drowsiness/Tiredness (General disorders) | 5 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 10 (17) | 8 (8)
GI upset (Gastrointestinal disorders) | 5 (5) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 17 (29) | 12 (20)
Upper respiratory infection (Infections and infestations) | 20 (31) | 14 (24)

LIMITATIONS AND CAVEATS:
Several secondary analyses. Subject non-compliance with eye tracking led to unreliable/uninterpretable data. Subjects and caregivers were unblinded at the time they completed the study. Limited number of girls in the study (total 9 girls).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No